CLINICAL TRIAL: NCT01350726
Title: Functional-three-dimensional Reconstruction and Functional Evaluation of Liver by 99MTc-GSA-SPECT Scintigraphy
Brief Title: Functional-three-dimensional Reconstruction of Liver by 99MTc-GSA-SPECT Scan
Acronym: GSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Dr. Yilei Mao, Peking Union Medical College Hospital
Other Study IDs: PUMCH-Liver surgery -GSA
Record Dates: First submitted 2011-05-08; First posted 2011-05-10 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Cirrhosis; Hepatic Carcinoma
Keywords: Cirrhosis; Hepatic Carcinoma
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal control: Subjects without liver cirrhosis and normal volunteers.
- Cirrhosis group: Subjects with liver cirrhosis.

SUMMARY:
The aims of this study were divided into three parts:

1. To develop a new software to carry out the functional-three- dimensional-reconstruction of the liver by 99mTc-GSA-SPECT scintigraphy
2. To probe a new dynamic model of the metabolism of the 99mTc-GSA.
3. To evaluate the liver function by 99mTc-GSA-SPECT scintigraphy before surgical treatment.

Study design:

1. Collectivity type: Prospective，randomized, controlled, multi-central clinical study.
2. Patients: The subjects were from different hospitals including: Peking Union Medical College Hospital (PUMCH).

Study arrangement:

This study was consisted of three parts:

ELIGIBILITY:
Inclusion Criteria:

* Patients that with benign tumor、hepatitis and hepatic carcinoma (with or without cirrhosis)diagnosed by examination of CT, ultrasound-B, and/or pathology.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects were from Peking Union Medical College Hospital from May, 2008 to the end of the study.
Sampling Method: Probability Sample
Enrollment: 0 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China